CLINICAL TRIAL: NCT02453893
Title: Double-blind,Double-simulation,Risperidone-controlled,Multicentre Clinical Trial of Iloperidone in Patients With Schizophrenia
Brief Title: Risperidone-controlled,Multicentre Clinical Trial of Iloperidone in Patients With Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPC-HC103/PRO/Ⅱ
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia
Keywords: Iloperidone; Risperidone; PANSS
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral iloperidone (Experimental): 2~12mg/day for 2 weeks,12~24mg/day for 6 weeks.
  Interventions: Drug: Iloperidone
- oral risperidone (Active Comparator): 1~3mg/day for 2 weeks,3~6mg/day for 6 weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Iloperidone
  Arms: oral iloperidone
Drug: Risperidone
  Arms: oral risperidone

SUMMARY:
This research is a Randomized, double-blind, risperidone-controlled, multicenter clinical study. Chinese subjects with Ischemic Schizophrenia.

DETAILED DESCRIPTION:
Subjects will randomly enter into one of two groups,the period of treatment is 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 to 65 years with schizophrenia;
* PANSS total score of at least 70 at screening and baseline;
* at least 2 more than 4 points in 7 of PANSS-P;
* informed consent.

Exclusion Criteria:

* allergy with iloperidone or risperidone;
* psychotic symptoms failing to improve after sufficient exposure to 2 antipsychotic treatment;
* any other primary Axis 1 psychiatric diagnosis;
* a history of alcohol or drug dependence in recent 1 year;
* at imminent risk of harm to self or others;
* systolic blood pressure≤90mmHg。

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the score of Positive and Negative syndrome scale to evaluation the severity of schizophrenia | 8 weeks

SECONDARY OUTCOMES:
the score of clinical global impressions to evaluation the severity of illness | 8 weeks
the score of clinical global impressions to evaluation the improvement of illness | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li hua fang, Ph.D, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China